CLINICAL TRIAL: NCT04778774
Title: Compare the Quadriceps Function of Adductor Canal Block Versus Femoral Nerve Block With Electromyography Following Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMUHIRB-F(I)-20200031
Record Dates: First submitted 2021-02-25; First posted 2021-03-03 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2021-02

CONDITIONS: Quadriceps Function Monitored With Electromyography
MeSH Terms: interventions — Nerve Block

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adductor canal block group (Experimental): Adductor canal block group
  Interventions: Procedure: Nerve block
- Femoral nerve block group (Experimental): Femoral nerve block group
  Interventions: Procedure: Nerve block

INTERVENTIONS:
Procedure: Nerve block — Two different nerve block types, Adductor canal block group and Femoral nerve block group

SUMMARY:
Adductor canal block and femoral nerve block are the most commonly used nerve blocks for pain control after total knee arthroplasty. The block area for adductor canal is a sensory branch near the knee area, which can potentially reduce the effect of motor blockage of quadriceps muscle. We try to proof adductor canal block can reduce the pain level after surgery effectively and preserve the muscle power of quadriceps muscle. Therefore, the rehabilitation course can be reduced and further lowering the risks of falling and complications.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 50 years old, not exceed 100 years old
* Diagnosed Primary Knee Osteoarthritis
* Accepted Total Knee Arthroplasty

Exclusion Criteria:

* Diagnosed Osteonecrosis
* Diagnosed inflammatory Arthritis、Rheumatoid Arthritis
* Accepted Revision Total Knee Arthroplasty
* Quadriceps muscle rupture, suture or repair history
* Neurological or orthopedic disorders that could affect quadriceps muscle power
* Allergy to amide anesthetics
* Patients who cannot obey or follow directions

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2021-10-18 (Actual); Study Completion 2021-11-29 (Actual)

PRIMARY OUTCOMES:
Quadriceps muscle Electromyography voltage level change before and after nerve block | compare difference of Quadriceps muscle Electromyography voltage level 12 weeks after surgery,data were measured post operation day 1, day 2, day 5, 2 weeks, 6 weeks and 12 weeks
  surface electromyography level

CONTACTS AND LOCATIONS:
Overall Officials: Hsuan-Ti Huang, M.D, Study Director — Kaohsiung Medical University
Locations (1):
- Kaohsiung Municipal Ta-Tung Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No